CLINICAL TRIAL: NCT00223067
Title: A Multi-Center Open-Labeled Study of the Administration of Allogenic and Autologous Regulatory Cells for the Induction of Donor-Specific Tolerance in Renal Allograft Recipients (Living Donor)
Brief Title: Induction of Donor-Specific Tolerance in Renal Allograft Recipients (Living Donor) With TAIZ-Monocytes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2004-04

CONDITIONS: Renal Transplantation
Keywords: renal transplantation; TAIZ

INTERVENTIONS:
Drug: TAIZ

SUMMARY:
reduce of immunsupression or introduce tolerance with so called TAIZ-monocytes in renal transplant patients

ELIGIBILITY:
Inclusion Criteria

Patients must meet all the following inclusion criteria to be considered for admission to the trial:

1. Male or female adult patients aged between 18 and 64 years (inclusive). A female of childbearing potential may be enrolled provided she:

   * has a negative pregnancy test at Screening and
   * is routinely using adequate contraception prior to and during the study and
   * agrees not to attempt to become pregnant during the study and
   * is not lactating A female of non-childbearing potential will be defined as one who has been postmenopausal for at least one year or has been surgically sterilised.
2. Patients receiving a first renal transplant.
3. Patients who fulfil the criteria to receive an allogenic renal transplant (according to the Eurotransplant (ET) manual on organ allocation and the Bundesärztekammer allocation criteria) and who are listed on a waiting list.
4. Patients who, after the nature of the study and the disclosure of their data has been explained to them, have freely given Informed Consent in writing.
5. In vitro demonstration of the suppressive effect of the donor TAIC for the donor-recipient pair.

Exclusion Criteria (for the recipient)

Exclusion Criteria (for the recipient):

Patients presenting any of the following exclusion criteria must not be included in the trial:

1. Patients who have received a renal transplant.
2. Patients who have an active infection at the time of entry into the study (Screening).
3. Recipient and donor pairs who show the following incompatible EBV or CMV constellation: the donor is EBV or CMV positive and the recipient is EBV or CMV negative.
4. Patients and/or donors who have positive evidence of HIV or have active virus hepatitis B and C.
5. Patients with a history of alcohol and/or drug abuse or sepsis.
6. Patients who are pregnant women or nursing mothers.
7. Known hypersensitivity or contraindication to one of the immunosuppressives administered during the course of the study: ATG, tacrolimus, or steroids (prednisolone).
8. Patients with a history or present symptoms of autoimmune vasculitis.
9. Detection of > 5% HLA antibodies (all current and historic values).
10. Patients with a malignancy or history of malignancy.
11. Patients with renal insufficiency due to a vasculitis.
12. Patients whose condition requires continuous systemic administration of immunosuppressives.
13. Missing immunosuppressive effect of the donor TAIC for the donor-recipient pair in vitro test.
14. Patients who are simultaneously participating or plan to participate in any other clinical study.
15. Psychiatric or emotional problems or lack of knowledge of the German language which would invalidate the giving of Informed Consent or limit the ability of the subject to comply with study requirements.
16. Unwillingness or inability to provide Informed Consent or to participate satisfactorily for the entire trial period
17. Patients with corresponding donors presenting any one of the exclusion criteria documented in the Eurotransplant guidelines ( ) must not be included in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-03; Study Completion 2006-05

PRIMARY OUTCOMES:
graft survival and reduction or withdrawal of immunosuppressives after treatment with Transplant-Acceptance Inducing Cells (TAIC) and autologous regulatory T cells (tregs)
serum creatinine
rejection episodes
necessity for re-introduction of any immunosuppressives.

SECONDARY OUTCOMES:
safety and tolerability of the treatment with Transplant-Acceptance Inducing Cells (TAIC) in terms of rejection episodes and Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Kunzendorf, MD, Principal Investigator — University of Schleswig-Holstein, Campus Kiel Department of Nephrology
Locations (1):
- University of Schleswig-Holstein, Campus Kiel, Department of Nephrology, Kiel, Germany